CLINICAL TRIAL: NCT03326570
Title: Comparative Effectiveness of Bronchoscopic Interventions for Malignant Airway Obstruction
Brief Title: Effectiveness of Bronchoscopic Interventions for Malignant Airway Obstruction
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-0563; NCI-2018-01276 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-10-20; First posted 2017-10-31 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Data collection post bronchoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bronchoscopy Data Collection: Medical information collected after bronchoscopy for up to 2 years.
  Interventions: Behavioral: Medical Data Collection

INTERVENTIONS:
Behavioral: Medical Data Collection — Medical information collected after bronchoscopy for up to 2 years.

SUMMARY:
The goal of this clinical research study is learn about side effects and the success of bronchoscopies when performed in cancer patients with and without symptoms.

This is an investigational study.

Up to 110 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, researchers will collect information from participant's medical records.

Length of Study:

Researchers will continue to collect participant's medical information for up to 2 years.

Additional Information:

Participant's data will be kept in a database on a password-protected computer in a secure office. This information will only be available to the study doctors and staff.

ELIGIBILITY:
Inclusion Criteria:

° All patients undergoing interventional bronchoscopy during the first 12 months will be enrolled, with follow-up occurring out to 2 years from the study startup (the duration of the grant).

Exclusion Criteria:

* Age less than 18 years,
* Inability to participate in telephone follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled for standard of care bronchoscopy at UT MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-08-25 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Time to Any Complication Requiring Treatment | 2 years
  Researchers will estimate the hazard function of time to any complications in the framework of competing risks while death is the competing risk.3 Researchers will graphically visualize the hazard function of time to any complications using Kernel smoothing method.

SECONDARY OUTCOMES:
Quality-Adjusted Survival | 2 years
  Researchers will evaluate the relationship between covariates and quality-adjusted survival.

OTHER OUTCOMES:
Early Intervention | 2 years
  Early intervention cases defined as those with anatomic narrowing and no or mild dyspnea (as measured by the Borg score).
Late Intervention | 2 years
  Late intervention cases defined as those with moderate or severe dyspnea due to airway narrowing.

CONTACTS AND LOCATIONS:
Overall Officials: David Ost, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ong P, Grosu HB, Debiane L, Casal RF, Eapen GA, Jimenez CA, Noor L, Ost DE. Long-term quality-adjusted survival following therapeutic bronchoscopy for malignant central airway obstruction. Thorax. 2019 Feb;74(2):141-156. doi: 10.1136/thoraxjnl-2018-211521. Epub 2018 Sep 25. PMID 30254139
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org